CLINICAL TRIAL: NCT01606150
Title: Lumbar Punctures in Neonates: Improving Success Rates and Minimizing Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left the insititution
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Courtney DeJesso, MD, Fellow, Georgetown University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MGUHNICULP
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-10

CONDITIONS: Meningitis
Keywords: neonate; late preterm; lumbar puncture; analgesia; pain; lidocaine
MeSH Terms: conditions — Meningitis; Agnosia; Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subcutaneous Lidocaine (Active Comparator): 0.1 ml/kg of 1% Lidocaine
  Interventions: Drug: 1% lidocaine
- Topical Lidocaine (Active Comparator): LMX-4, 1 gram placed over lumbar puncture needle insertion site 30 minutes prior to the procedure
  Interventions: Drug: topical lidocaine

INTERVENTIONS:
Drug: 1% lidocaine — 0.1 ml/kg of 1% lidocaine injected over lumbar puncture needle insertion site 2 minutes prior to procedure
  Other Names: LIDOCAINE
  Arms: Subcutaneous Lidocaine
Drug: topical lidocaine — 1 gram placed over lumbar puncture needle insertion point 30 minutes prior to procedure
  Other Names: LMX-4
  Arms: Topical Lidocaine

SUMMARY:
The purpose of this study is to compare two medications used to numb an infant's back when performing a lumbar puncture. A lumbar puncture (LP) is often needed in newborns to obtain cerebrospinal fluid (CSF). This is achieved by inserting a small needle between the infant's vertebrae. In the past, doctors did not know if newborns could feel the pain from a procedure like this in the same way that adults do. Investigators now know that the newborns do experience pain during this procedure, but we do not know the best way to control this pain. Investigators also think that when the newborns have pain, they move during the test. The movement can increase the chance of having blood mix with this normally clear fluid leading to limitations in our clinical application of these results. This study will compare the injected and topical forms of Lidocaine to see which gives us better pain control and more clear results. The investigators hypothesize that subcutaneous 1% Lidocaine, due to its deeper penetration, will be 25% superior to topical liposomal Lidocaine (LMX-4) in both the rate of clinically useful results and pain scores. The investigators hypothesize that both forms of Lidocaine will be 25% superior to our historical control cohort in the rate of clinically useful results.

DETAILED DESCRIPTION:
When the decision is made that an infant needs a lumbar puncture for clinical indications, parental consent will be obtained for the actual procedure and a separate consent for participation in this study will be attached. Randomization for this study will be via permuted block randomization. The expected 122 patients will be pre-randomized, with the arm for each patient number 1 through 122 sealed in an envelope. After consent is obtained the patient will be assigned the next numerical study identification number and the corresponding envelope will be opened. If the infant has been randomized to the topical liposomal lidocaine group, 1 gram of LMX-4 will be placed over the L3-L4 space immediately, covered with a cotton ball and occlusive tegaderm, for minimum 30 minutes prior to the needle insertion during the lumbar puncture (LP). While the LMX-4 is in place, other procedures that are part of a routine septic work-up may be performed. Thus, the application of this medication should not cause an unnecessary delay in the ultimate procedure or antibiotic administration.

If the infant has been randomized to the subcutaneous lidocaine group, after using sterile procedure to prepare the area, 0.1ml/kg of 1% Lidocaine will be injected using a 25 gauge tuberculin needle over the L3-L4 region. The injection point will be below the actual level desired with the needle going in at a 5-10 degree angle and moving toward the head after insertion. A subcutaneous wheal will form over the desired L3-L4 space when the Lidocaine is injected. The provider will wait at minimum 2 minutes after the injection of the Lidocaine prior to the insertion of the LP needle. Once the required time for local anesthesia in either arm has elapsed, the procedure will be performed with routine technique.

With consent for the video portion of the study, a video camera will be set up to tape the infants face only during the procedure with notation of the LP needle insertion(s). During the procedure, an assistant will record heart rate and oxygen saturation values. The information from the video and documented vital signs will be used to assign a PIPP score by a blinded investigator. Once the procedure is complete the following information will be obtained for study purposes, in addition to the above video tape and vital signs: infant gestational age, infant birth weight, gender, day of life of procedure, level of provider(s) performing the procedure, attempts required to obtain cerebrospinal fluid (CSF) specimen, color of fluid (clear, pink, xanthochromic, or grossly bloody), presence of CSF culture, and Red Blood Cell count of CSF specimen. Infants in our institution will already be monitored continuously and will continue to be so for at minimum 6 hours after the procedure. Any adverse reaction that could be attributed to the procedure or medications used for the procedure will be recorded, with the most expected reaction to be a skin rash. Additional changes in the infant, such as apnea, sustained arrhythmia, oxygen desaturation 10% below baseline, or seizure will also be noted whether or not it is thought to be associated with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* neonate requiring lumbar puncture
* gestational age at birth equal to or greater than 34 weeks

Exclusion Criteria:

* on mechanical ventilation
* receiving sedation (opioids or benzodiazepines)
* suspected congenital spinal anomaly
* infants older than 1 week of life

Max Age: 8 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith J PALAFOUTAS, RN, Study Director — Georgetown University Hospital
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
THERE IS NO DATA TO SHARE

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subcutaneous Lidocaine | Topical Lidocaine
Started | 0 | 0
Completed | 0 (Enrollment was only for two months in 2012 due to technical and enrollment problems) | 0 (Enrollment was only for two months in 2012 due to technical and enrollment problems)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subcutaneous Lidocaine | Topical Lidocaine | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
Age, Continuous [Mean (Standard Deviation); unit: years]
Sex: Female, Male [Count of Participants; unit: Participants]
Race (NIH/OMB) [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Lumbar Puncture Success Rate
Description: Success defined as cerebrospinal fluid for a culture and red blood cell count less than 1000
Time Frame: immediately following the procedure
Arm/Group | Subcutaneous Lidocaine | Topical Lidocaine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Premature Infant Pain Profile (PIPP) Score
Description: PIPP score assigned by a blinded outcome assessor by viewing video tapes of the infant's face during the procedure and vital sign changes during that time frame
Time Frame: data collected during the procedure, PIPP score assigned within one month by viewing collected data
Arm/Group | Subcutaneous Lidocaine | Topical Lidocaine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Subcutaneous Lidocaine | Topical Lidocaine
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study proved to be very difficult to execute in a busy NICU due to clinical practice biases and technical difficulties in establishing masked treatment. The Investigator left the Fellowship program before any results could be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No